CLINICAL TRIAL: NCT00849836
Title: The Study for The Identification of Novel Biomarkers in Chronic Airway Inflammatory Disorders
Brief Title: Novel Biomarkers in Chronic Airway Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chonbuk National University (Other)
Responsible Party: Yong Chul Lee, Chonbuk National University Medical School
Other Study IDs: RCPD
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Acute exacerbation
- Stable disease
- Healthy control

SUMMARY:
The purpose of this study is:

* To define The differences of bio-chemical phenotypes in chronic airway inflammatory diseases.
* To identify novel biomarkers in chronic airway inflammatory diseases as a screening, diagnostic, or monitoring marker.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years olds
* Both sexes
* Asthma or COPD was diagnosed according to the criteria of the American Thoracic Society, GINA, GOLD guideline
* Acute exacerbation was defined by the criteria of the American Thoracic Society, GINA, GOLD guideline
* For stable disease, none of the subjects had received inhaled or oral corticosteroids or any other anti-inflammatory drugs, had an exacerbation history in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute exacerbation of asthma or COPD, patients with stable status of those disease, and the healthy control subjects
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Medical School, Jeonju, South Korea